CLINICAL TRIAL: NCT07224061
Title: Promoting Asthma Guidelines and Management Through Technology-Based Intervention and Care Coordination in Clinics and Schools (PRAGMATIC-S)
Brief Title: Promoting Asthma Management Guidelines With Technology-Based Intervention and Care Coordination in Clinics and Schools
Acronym: PRAGMATIC-S
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-17054; R01HL181061 (NIH)
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Asthma in Children

STUDY DESIGN:
Intervention Model Description: Cluster randomized design. Prior to participant enrollment, each practice will be matched into 9 pairs based on size of the practice and provider type. Practices will then be randomly selected within each pair to receive PRAGMATIC-S or remain as an Enhanced Usual Care (eUC) site. Practices will join study in 5 waves (2-4 practices per wave).
Masking Description: Follow up assessments will be collected by blinded interviewers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRAGMATIC-S (Experimental): Primary Care Providers (PCPs) will use guideline-based prompts within EHR; PCPs and caregivers will complete medication administration forms electronically with forms routed directly to schools to receive asthma medications at the school, and asthma outreach workers will serve as liaison between families, PCPs, schools and provide care coordination and support.
  Interventions: Behavioral: PRAGMATIC-S
- Enhanced Usual Care (No Intervention): Standard of care EHR clinician prompts for guideline-based asthma care

INTERVENTIONS:
Behavioral: PRAGMATIC-S — Intervention combines EHR-based guideline prompts, electronic MAF submission, school-based directly observed therapy (DOT), and Asthma Outreach Workers (AOWs) providing care coordination, adherence support, and communication between families, schools, and providers.
  Arms: PRAGMATIC-S

SUMMARY:
The overall goal of this research study is to evaluate a multi-level program called PRAGMATIC-S to improve the delivery of guideline-based asthma care through a unique partnership between clinical practices and schools. PRAGMATIC-S represents a novel approach that addresses multiple barriers to adherence by bridging primary care and schools, ensuring delivery of guideline-based asthma care to urban children across these settings thereby improving adherence to therapy and clinical outcomes.

DETAILED DESCRIPTION:
The research team will conduct a cluster randomized controlled trial, enrolling 420 children, ages 4-12, from 18 Montefiore clinics during office visits. Children in the intervention group (PRAGMATIC-S) will receive updated guideline-based care prompts, with providers completing the medication administration form (MAF), electronically signing it, and routing it directly to the school via the EHR system. Asthma Outreach Worker (AOW) care coordination will support daily adherence to prescribed treatments at home and school. Children in the control group will receive enhanced usual care, which includes EHR prompts for guideline-based care but without the additional PRAGMATIC-S components.

Participants will be followed for 12 months. Outcomes will be assessed as outlined in this registration.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma documented in EHR
* Persistent or uncontrolled asthma, defined by age-specific guidelines (symptoms ≥2 days/week, rescue medication use ≥2 days/week, nighttime symptoms ≥2 days/month, or ≥2 steroid-requiring episodes/year)
* Age 4 to 12 years, attending pre-kindergarten through 6th grade in NYC public schools
* Caregiver able to speak English or Spanish
* Consent from primary caregiver and assent from child (if ≥7 years)
* Presence of phone and device (smartphone, iPad, or computer) to complete electronic forms

Exclusion Criteria:

* Family plans to leave school/city within 6 months
* Significant comorbidities (e.g., congenital heart disease, cystic fibrosis, chronic lung disease)
* Children in foster care or situations where legal guardian consent cannot be obtained
* Participation in concurrent asthma intervention study
* Severe developmental delay precluding completion of ACT questionnaire

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Asthma Control - continuous | Baseline, 4 months, 8 months, and 12 months
  Asthma control will be measured using the Childhood Asthma Control Test (cACT), 7-item scale which determines a score based on the sum of the response codes. The child answers the first 4 questions on a 4-point scale ranging from 0-3 and the caregiver provides responses for the final 3 items using a reverse-coded scale ranging from 0-5, yielding an overall possible scoring range of 0-27, with higher scores indicating better asthma control.
  Asthma control will be analyzed as a continuous variable.

SECONDARY OUTCOMES:
Pediatric Asthma Caregiver's Quality of Life | Baseline, 4 months, 8 months, and 12 months
  The caregiver's quality of life will be assessed using the validated Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ; also referred to as Juniper's Asthma Quality of Life Questionnaire). This questionnaire consists of 13 items which evaluate the impact of the child's asthma on the caregiver's quality of life. Responses to each item are rated on a 7-point scale ranging from 1-7, wherein 1 means "all of the time" or "very, very worried/concerned," and 7 means "none of the time" or "not worried/concerned," yielding an overall possible scoring range of 7-91, such that higher scores are indicative of less asthma related quality of life impairment.
Percent of participants with 1 or more guideline-based corrective actions taken | Up to 24 months (following intervention)
  Percent of participants with 1 or more guideline-based corrective actions taken (i.e., controller medication prescription or adjustment, trigger evaluation), as recorded in the electronic health record (EHR), will be summarized by study arm.
Asthma Control - dichotomous | Baseline, 4 months, 8 months, and 12 months
  Asthma control will also be measured as a dichotomous variable using the Childhood Asthma Control Test (cACT), 7-item scale which determines a score based on the sum of the response codes. The child answers the first 4 questions on a 4-point scale ranging from 0-3 and the caregiver provides responses for the final 3 items using a reverse-coded scale ranging from 0-5, yielding an overall possible scoring range of 0-27, with higher scores indicating better asthma control.
  Asthma control will be analyzed as dichotomous variable with a score of 19 or less indicating uncontrolled asthma.

OTHER OUTCOMES:
Health care utilization - number of Emergency Department (ED) visits for asthma | every 4 months up to 12 months
  The number of ED visits directly related to asthma will be summarized by study arm every four months up to 12 months in total.
Health care utilization - number of hospitalizations for asthma | every 4 months up to 12 months
  The number of hospitalizations directly related to asthma will be summarized by study arm every four months up to 12 months in total.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Reznik, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Children's Hospital at Montefiore, Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Walters S, Wilson L, Konty K, Day S, Agerton T, Olson C. Disparities among children with asthma in New York City. Epi Data Brief (126); September 2021.
- [Background] Black LI, Benson V. Tables of Summary Health Statistics for U.S. Children: 2018 National Health Interview Survey.
- [Background] Reznik M, Jaramillo Y, Wylie-Rosett J. Demonstrating and assessing metered-dose inhaler-spacer technique: pediatric care providers' self-reported practices and perceived barriers. Clin Pediatr (Phila). 2014 Mar;53(3):270-6. doi: 10.1177/0009922813512521. Epub 2013 Dec 12. PMID 24336438
- [Background] Frey SM, Fagnano M, Halterman JS. Caregiver education to promote appropriate use of preventive asthma medications: what is happening in primary care? J Asthma. 2016;53(2):213-9. doi: 10.3109/02770903.2015.1075549. Epub 2015 Aug 18. PMID 26288255
- [Background] Halterman JS, Auinger P, Conn KM, Lynch K, Yoos HL, Szilagyi PG. Inadequate therapy and poor symptom control among children with asthma: findings from a multistate sample. Ambul Pediatr. 2007 Mar-Apr;7(2):153-9. doi: 10.1016/j.ambp.2006.11.007. PMID 17368410
- [Background] Okelo SO, Siberry GK, Solomon BS, Bilderback AL, Yamazaki M, Hetzler T, Ferrell CL, Dhepyasuwan N, Serwint JR; CORNET Investigators. Asthma treatment decisions by pediatric residents do not consistently conform to guidelines or improve with level of training. Acad Pediatr. 2014 May-Jun;14(3):287-93. doi: 10.1016/j.acap.2013.12.008. Epub 2014 Mar 12. PMID 24629404
- [Background] National Heart Lung and Blood Institute. National Asthma Education and Prevention Program. Expert panel report 3: guidelines for the diagnosis and management of asthma. NIH Publication Number 08-5846. Bethesda, MD: 2007.
- [Background] Liu AH, Zeiger R, Sorkness C, Mahr T, Ostrom N, Burgess S, Rosenzweig JC, Manjunath R. Development and cross-sectional validation of the Childhood Asthma Control Test. J Allergy Clin Immunol. 2007 Apr;119(4):817-25. doi: 10.1016/j.jaci.2006.12.662. Epub 2007 Mar 13. PMID 17353040
- [Background] Schatz M, Zeiger RS, Drane A, Harden K, Cibildak A, Oosterman JE, Kosinski M. Reliability and predictive validity of the Asthma Control Test administered by telephone calls using speech recognition technology. J Allergy Clin Immunol. 2007 Feb;119(2):336-43. doi: 10.1016/j.jaci.2006.08.042. Epub 2006 Dec 27. PMID 17194469
- [Background] Halterman JS, Borrelli B, Fisher S, Szilagyi P, Yoos L. Improving care for urban children with asthma: design and methods of the School-Based Asthma Therapy (SBAT) trial. J Asthma. 2008 May;45(4):279-86. doi: 10.1080/02770900701854908. PMID 18446591
- [Background] Halterman JS, Szilagyi PG, Fisher SG, Fagnano M, Tremblay P, Conn KM, Wang H, Borrelli B. Randomized controlled trial to improve care for urban children with asthma: results of the School-Based Asthma Therapy trial. Arch Pediatr Adolesc Med. 2011 Mar;165(3):262-8. doi: 10.1001/archpediatrics.2011.1. PMID 21383275
- [Background] Halterman JS, Fagnano M, Montes G, Fisher S, Tremblay P, Tajon R, Sauer J, Butz A. The school-based preventive asthma care trial: results of a pilot study. J Pediatr. 2012 Dec;161(6):1109-15. doi: 10.1016/j.jpeds.2012.05.059. Epub 2012 Jul 10. PMID 22785264
- [Background] Halterman JS, Fagnano M, Tajon RS, Tremblay P, Wang H, Butz A, Perry TT, McConnochie KM. Effect of the School-Based Telemedicine Enhanced Asthma Management (SB-TEAM) Program on Asthma Morbidity: A Randomized Clinical Trial. JAMA Pediatr. 2018 Mar 5;172(3):e174938. doi: 10.1001/jamapediatrics.2017.4938. Epub 2018 Mar 5. PMID 29309483
- [Background] Halterman JS, Riekert KA, Fagnano M, Tremblay PJ, Blaakman SW, Tajon R, Wang H, Borrelli B. Effect of the School-Based Asthma Care for Teens (SB-ACT) program on asthma morbidity: a 3-arm randomized controlled trial. J Asthma. 2022 Mar;59(3):494-506. doi: 10.1080/02770903.2020.1856869. Epub 2021 Jan 8. PMID 33307900
- [Background] Cain A, Reznik M. The Principal and Nurse Perspective on Gaps in Asthma Care and Barriers to Physical Activity in New York City Schools: A Qualitative Study. Health Educ Behav. 2018 Jun;45(3):410-422. doi: 10.1177/1090198117736351. Epub 2017 Oct 31. PMID 29084455
- [Background] Reznik M, Bauman LJ, Okelo SO, Halterman JS. Asthma identification and medication administration forms in New York City schools. Ann Allergy Asthma Immunol. 2015 Jan;114(1):67-68.e1. doi: 10.1016/j.anai.2014.10.006. Epub 2014 Oct 24. No abstract available. PMID 25454012
- [Background] Reznik M, Halterman JS. School asthma policies and teachers' confidence and attitudes about their role in asthma management. Ann Allergy Asthma Immunol. 2016 May;116(5):473-5. doi: 10.1016/j.anai.2016.03.005. Epub 2016 Mar 22. No abstract available. PMID 27013055
- [Background] Expert Panel Working Group of the National Heart, Lung, and Blood Institute (NHLBI) administered and coordinated National Asthma Education and Prevention Program Coordinating Committee (NAEPPCC); Cloutier MM, Baptist AP, Blake KV, Brooks EG, Bryant-Stephens T, DiMango E, Dixon AE, Elward KS, Hartert T, Krishnan JA, Lemanske RF Jr, Ouellette DR, Pace WD, Schatz M, Skolnik NS, Stout JW, Teach SJ, Umscheid CA, Walsh CG. 2020 Focused Updates to the Asthma Management Guidelines: A Report from the National Asthma Education and Prevention Program Coordinating Committee Expert Panel Working Group. J Allergy Clin Immunol. 2020 Dec;146(6):1217-1270. doi: 10.1016/j.jaci.2020.10.003. PMID 33280709
- [Background] Hsia BC, Singh AK, Njeze O, Cosar E, Mowrey WB, Feldman J, Reznik M, Jariwala SP. Developing and evaluating ASTHMAXcel adventures: A novel gamified mobile application for pediatric patients with asthma. Ann Allergy Asthma Immunol. 2020 Nov;125(5):581-588. doi: 10.1016/j.anai.2020.07.018. Epub 2020 Jul 22. PMID 32711031
- [Background] Hsia BC, Wu S, Mowrey WB, Jariwala SP. Evaluating the ASTHMAXcel Mobile Application Regarding Asthma Knowledge and Clinical Outcomes. Respir Care. 2020 Aug;65(8):1112-1119. doi: 10.4187/respcare.07550. Epub 2020 Jun 2. PMID 32487751
- [Background] Halterman JS, Tajon R, Tremblay P, Fagnano M, Butz A, Perry TT, McConnochie KM. Development of School-Based Asthma Management Programs in Rochester, New York: Presented in Honor of Dr Robert Haggerty. Acad Pediatr. 2017 Aug;17(6):595-599. doi: 10.1016/j.acap.2017.04.008. Epub 2017 Apr 18. PMID 28434913
- [Background] Juniper EF, Guyatt GH, Feeny DH, Ferrie PJ, Griffith LE, Townsend M. Measuring quality of life in the parents of children with asthma. Qual Life Res. 1996 Feb;5(1):27-34. doi: 10.1007/BF00435966. PMID 8901364
- [Background] Taminskiene V, Alasevicius T, Valiulis A, Vaitkaitiene E, Stukas R, Hadjipanayis A, Turner S, Valiulis A. Quality of life of the family of children with asthma is not related to asthma severity. Eur J Pediatr. 2019 Mar;178(3):369-376. doi: 10.1007/s00431-018-3306-8. Epub 2019 Jan 4. PMID 30607508
- [Background] Smith T, Mills K, Cober MP, Fenn NE 3rd, Hill C, King M, Pauley JL, Eiland L, Sierra C, Omecene NE. Updates in the treatment of asthma in pediatrics: A review for pharmacists. Am J Health Syst Pharm. 2024 Apr 19;81(9):e210-e219. doi: 10.1093/ajhp/zxad326. PMID 38146826
- [Background] Hogan A, Kyler K, Seguin C. 2022. Get SMART: Implementation of Updated Asthma Guidelines for Pediatric Hospitalists.
- [Background] Beasley R, Harper J, Bird G, Maijers I, Weatherall M, Pavord ID. Inhaled Corticosteroid Therapy in Adult Asthma. Time for a New Therapeutic Dose Terminology. Am J Respir Crit Care Med. 2019 Jun 15;199(12):1471-1477. doi: 10.1164/rccm.201810-1868CI. PMID 30645143
- [Background] Bender B, Wamboldt FS, O'Connor SL, Rand C, Szefler S, Milgrom H, Wamboldt MZ. Measurement of children's asthma medication adherence by self report, mother report, canister weight, and Doser CT. Ann Allergy Asthma Immunol. 2000 Nov;85(5):416-21. doi: 10.1016/s1081-1206(10)62557-4. PMID 11101187
- [Background] O'Connor SL, Bender BG, Gavin-Devitt LA, Wamboldt MZ, Milgrom H, Szefler S, Rand C, Wamboldt FS. Measuring adherence with the Doser CT in children with asthma. J Asthma. 2004 Sep;41(6):663-70. doi: 10.1081/jas-200026434. PMID 15584316
- [Background] Mosnaim G, Li H, Martin M, Richardson D, Belice PJ, Avery E, Ryan N, Bender B, Powell L. The impact of peer support and mp3 messaging on adherence to inhaled corticosteroids in minority adolescents with asthma: a randomized, controlled trial. J Allergy Clin Immunol Pract. 2013 Sep-Oct;1(5):485-93. doi: 10.1016/j.jaip.2013.06.010. Epub 2013 Aug 30. PMID 24565620
- [Background] Makhecha S, Chan A, Pearce C, Jamalzadeh A, Fleming L. Novel electronic adherence monitoring devices in children with asthma: a mixed-methods study. BMJ Open Respir Res. 2020 Nov;7(1):e000589. doi: 10.1136/bmjresp-2020-000589. PMID 33154086
- [Background] LaForce C, Albers FC, Cooper M, Danilewicz A, Dunsire L, Rees R, Cappelletti C. A Fully Decentralized Randomized Controlled Study of As-Needed Albuterol-Budesonide Fixed-Dose Inhaler in Mild Asthma: The BATURA Study Design. J Asthma Allergy. 2024 Aug 23;17:801-811. doi: 10.2147/JAA.S471134. eCollection 2024. PMID 39193207
- [Background] Krings JG, Wojcik KM, Chen V, Sekhar TC, Harris K, Zulich A, Sumino K, Brownson R, Lenze E, Castro M. Symptom-driven inhaled corticosteroid/long-acting beta-agonist therapy for adult patients with asthma who are non-adherent to daily maintenance inhalers: a study protocol for a pragmatic randomized controlled trial. Trials. 2022 Dec 5;23(1):975. doi: 10.1186/s13063-022-06916-3. PMID 36471430
- [Background] Sun Y, Jariwala S, Reznik M. Measurement of adherence to inhaled corticosteroids by self-report and electronic medication monitoring. J Asthma. 2023 Jul;60(7):1299-1305. doi: 10.1080/02770903.2022.2144352. Epub 2022 Dec 1. PMID 36343353
- [Background] Cohen JL, Mann DM, Wisnivesky JP, Home R, Leventhal H, Musumeci-Szabo TJ, Halm EA. Assessing the validity of self-reported medication adherence among inner-city asthmatic adults: the Medication Adherence Report Scale for Asthma. Ann Allergy Asthma Immunol. 2009 Oct;103(4):325-31. doi: 10.1016/s1081-1206(10)60532-7. PMID 19852197
- [Background] Williams LK, Joseph CL, Peterson EL, Wells K, Wang M, Chowdhry VK, Walsh M, Campbell J, Rand CS, Apter AJ, Lanfear DE, Tunceli K, Pladevall M. Patients with asthma who do not fill their inhaled corticosteroids: a study of primary nonadherence. J Allergy Clin Immunol. 2007 Nov;120(5):1153-9. doi: 10.1016/j.jaci.2007.08.020. Epub 2007 Oct 22. PMID 17936894
- [Background] Apter AJ, Wan F, Reisine S, Bender B, Rand C, Bogen DK, Bennett IM, Bryant-Stephens T, Roy J, Gonzalez R, Priolo C, Have TT, Morales KH. The association of health literacy with adherence and outcomes in moderate-severe asthma. J Allergy Clin Immunol. 2013 Aug;132(2):321-7. doi: 10.1016/j.jaci.2013.02.014. Epub 2013 Apr 13. PMID 23591273
- [Background] De Keyser HEH, Kaye L, Anderson WC, Gondalia R, Theye B, Szefler SJ, Stempel DA. Electronic medication monitors help determine adherence subgroups in asthma. Respir Med. 2020 Apr;164:105914. doi: 10.1016/j.rmed.2020.105914. Epub 2020 Feb 19. PMID 32094102
- [Background] Julius SM, Sherman JM, Hendeles L. Accuracy of three electronic monitors for metered-dose inhalers. Chest. 2002 Mar;121(3):871-6. doi: 10.1378/chest.121.3.871. PMID 11888975
- [Background] Loucks J, Zuckerman AD, Berni A, Saulles A, Thomas G, Alonzo A. Proportion of days covered as a measure of medication adherence. Am J Health Syst Pharm. 2022 Mar 7;79(6):492-496. doi: 10.1093/ajhp/zxab392. No abstract available. PMID 34637496
- [Background] Horne R. Compliance, adherence, and concordance: implications for asthma treatment. Chest. 2006 Jul;130(1 Suppl):65S-72S. doi: 10.1378/chest.130.1_suppl.65S. PMID 16840369
- [Background] Reznik M, Silver EJ, Cao Y. Evaluation of MDI-spacer utilization and technique in caregivers of urban minority children with persistent asthma. J Asthma. 2014 Mar;51(2):149-54. doi: 10.3109/02770903.2013.854379. Epub 2013 Oct 22. PMID 24131031
- [Background] Interiano B, Guntupalli KK. Metered-dose inhalers. Do health care providers know what to teach? Arch Intern Med. 1993 Jan 11;153(1):81-5. doi: 10.1001/archinte.153.1.81. PMID 8422202
- [Background] Manzella BA, Brooks CM, Richards JM Jr, Windsor RA, Soong S, Bailey WC. Assessing the use of metered dose inhalers by adults with asthma. J Asthma. 1989;26(4):223-30. doi: 10.3109/02770908909073253. PMID 2702229
- [Background] O'Connor KS, Osborn L, Olson L, Blumberg SJ, Frankel MR, Srinath KP, Giambo P. Design and operation of the National Asthma Survey. Vital Health Stat 1. 2008 Aug;(46):1-122. PMID 18958992
- [Background] Horne R, Weinman J, Hankins M. The beliefs about medicines questionnaire: the development and evaluation of a new method for assessing the cognitive representation of medication. Psychol Health. 1999;14:1-24.
- [Background] Horne R. Patients' beliefs about treatment: the hidden determinant of treatment outcome? J Psychosom Res. 1999 Dec;47(6):491-5. doi: 10.1016/s0022-3999(99)00058-6. No abstract available. PMID 10661596
- [Background] Sidora-Arcoleo K, Feldman J, Serebrisky D, Spray A. Validation of the Asthma Illness Representation Scale (AIRS). J Asthma. 2010 Feb;47(1):33-40. doi: 10.3109/02770900903362668. PMID 20100018
- [Background] Sidora-Arcoleo KJ, Feldman J, Serebrisky D, Spray A. Validation of the Asthma Illness Representation Scale-Spanish (AIRS-S). J Asthma. 2010 May;47(4):417-21. doi: 10.3109/02770901003702832. PMID 20528596
- [Background] Kan K, Fierstein J, Boon K, Madeleine Kanaley, Zavos P, Volerman A, Vojta D, Gupta RS. Parental quality of life and self-efficacy in pediatric asthma. J Asthma. 2021 Jun;58(6):742-749. doi: 10.1080/02770903.2020.1731825. Epub 2020 Feb 25. PMID 32072838
- [Background] Bursch B, Schwankovsky L, Gilbert J, Zeiger R. Construction and validation of four childhood asthma self-management scales: parent barriers, child and parent self-efficacy, and parent belief in treatment efficacy. J Asthma. 1999;36(1):115-28. doi: 10.3109/02770909909065155. PMID 10077141
- [Background] Fiese BH, Wamboldt FS, Anbar RD. Family asthma management routines: connections to medical adherence and quality of life. J Pediatr. 2005 Feb;146(2):171-6. doi: 10.1016/j.jpeds.2004.08.083. PMID 15689901
- [Background] Clark NM, Gong M, Schork MA, Maiman LA, Evans D, Hurwitz ME, Roloff D, Mellins RB. A scale for Assessing Health Care Providers' Teaching and Communication Behavior regarding asthma. Health Educ Behav. 1997 Apr;24(2):245-56. doi: 10.1177/109019819702400211. PMID 9079582
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Matt GE, Wahlgren DR, Hovell MF, Zakarian JM, Bernert JT, Meltzer SB, Pirkle JL, Caudill S. Measuring environmental tobacco smoke exposure in infants and young children through urine cotinine and memory-based parental reports: empirical findings and discussion. Tob Control. 1999 Autumn;8(3):282-9. doi: 10.1136/tc.8.3.282. PMID 10599573
- [Background] Holm, S. A simple sequentially rejective multiple test procedure. Scandinavian Journal of Statistics. 1979; 6 (2): 65-70.
- [Background] Liang, K.Y. and Zeger, S. L. (1986), Longitudinal Data Analysis Using Generalized Linear Models. Biometrika, Vol. 73, No. 1., pp. 13-22.
- [Background] Rubin, D.B. Inference and missing data. Biometrika, 1976:63, 581-592.
- [Background] Imai K, Keele L, Tingley D. A general approach to causal mediation analysis. Psychol Methods. 2010 Dec;15(4):309-34. doi: 10.1037/a0020761. PMID 20954780